CLINICAL TRIAL: NCT06454240
Title: A Randomized Phase 2, Double-blind, Placebo-controlled, Parallel-group, 2-arm Study to Assess the Efficacy, Safety, and Tolerability of Subcutaneous Lunsekimig in Adult Participants With Chronic Rhinosinusitis With Nasal Polyps (CRSwNP)
Brief Title: A Proof-of-concept Study of Lunsekimig Compared With Placebo in Adults With Chronic Rhinosinusitis With Nasal Polyps
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACT18207; 2024-511261-11 (Registry Identifier: CTIS); U1111-1300-6978 (Other: ICTRP)
Record Dates: First submitted 2024-06-06; First posted 2024-06-12 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Chronic Rhinosinusitis With Nasal Polyps

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Placebo Comparator): Participant will receive placebo subcutaneous (SC) every 4 weeks and intranasal mometasone furoate nasal spray (MFNS) for 24 weeks.
  Interventions: Drug: placebo
- Arm 2 (Experimental): Participant will receive lunsekimig subcutaneous (SC) every 4 weeks and intranasal mometasone furoate nasal spray (MFNS) for 24 weeks.
  Interventions: Drug: lunsekimig

INTERVENTIONS:
Drug: lunsekimig — Pharmaceutical form:solution for injection-Route of administration:subcutaneous
  Other Names: SAR443765
  Arms: Arm 2
Drug: placebo — Pharmaceutical form:solution for injection-Route of administration:subcutaneous
  Arms: Arm 1

SUMMARY:
This is a parallel, Phase 2, 2-arm, multicenter, randomized, double-blind, placebo-controlled, proof-of-concept study for treatment of CRSwNP.

The purpose of this study is to assess the efficacy, safety, and tolerability of add-on therapy with subcutaneous lunsekimig in adult participants (aged 18 to 70 years, inclusive) with CRSwNP who are inadequately controlled on intranasal corticosteroid treatment. Participants with and without co-morbid asthma will be included in the study, and lung function will be assessed in both groups.

The study duration will be up to approximately 40 weeks per participant, including 4 weeks of screening run-in period, 24 weeks of intervention period, and 12 weeks of follow-up.

ELIGIBILITY:
Inclusion Criteria:

- A minimum bilateral nasal polyp score of 5 out of a maximum score of 8 for both nostrils (with at least a score of 2 for each nostril) despite use of intranasal corticosteroid treatment for at least 2 months prior to screening

Ongoing symptoms for at least 2 months prior to screening, including:

* Nasal congestion, blockage, or obstruction with moderate or severe symptom severity at screening (Score 2 or 3 on NC Score) and a weekly average severity score of at least 1 (range 0 to 3) at randomization (NC Score: 0=no symptoms, 1=mild, 2=moderate, and 3=severe).
* At least 1 of the following 2 symptoms: (1) partial loss of smell (hyposmia) or total loss of smell (anosmia); (2) anterior and/or posterior rhinorrhea.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

* Patient who has received any therapies such as for example systemic corticosteroids, anti-IgE therapy, monoclonal antibody and some others in the specified timeframe(s) prior to the screening visit
* Patients who have undergone any nasal/sinus surgery within 6 months before screening or for whom NPS cannot be determined accurately on endoscopy due to anatomic changes to the nasal cavity from past nasal/sinus surgery
* Patients with conditions/concomitant diseases making them non evaluable for the primary efficacy endpoint
* Signs or a CT scan suggestive of Allergic fungal rhinosinusitis
* Active/chronic helminthic infection
* History of human immunodeficiency virus (HIV) infection or positive HIV screen (Anti-HIV- and HIV-2 antibodies) at screening visit
* Patients with positive or indeterminate hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb), or hepatitis C antibody at screening visit NOTE: The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2024-07-17 (Actual); Primary Completion 2026-01-29 (Actual); Study Completion 2026-04-23 (Estimated)

PRIMARY OUTCOMES:
Change in bilateral endoscopic nasal polyp score (NPS). | From baseline to Week 24
  This score (NPS) is the sum of the right and left nostril scores, as evaluated by means of nasal endoscopy. NP is graded based on polyp size where: 0- no polyps and 4- large polyps causing complete obstruction of the inferior nasal cavity.

SECONDARY OUTCOMES:
Change in patient-reported nasal congestion/obstruction score | From baseline to Week 24
  Patient-reported nasal congestion/obstruction score. Score is using a 0-3 categorical scale where 0 = no symptoms, 1 = mild symptoms, 2 = moderate symptoms and 3 = severe symptoms
Change in Lund-Mackay CT score | From baseline to Week 24
  Lund-Mackay system is based on scoring bilateral areas of opacification with points given for degree of sinus opacification in each reagion: 0 = normal, 1 = partial opacification, 2 = total opacification.
Change in the percent of maxillary sinus volume occupied by disease on CT scan. | From baseline to Week 24
Change in SNOT-22 total score. | From baseline to Week 24
  The SNOT-22 is a 22-item health-related outcomes assessment. The 22-question SNOT-22 is scored as 0 (no problem) to 5 (problem as bad as it can be) with a total range from 0 to 110 (higher scores indicate poorer outcomes).
Change in patient-reported total symptom score (nasal congestion/obstruction, anterior or posterior rhinorrhea, and loss of smell). | From baseline to Week 24
  Score is using a 0-3 categorical scale where 0 = no symptoms, 1 = mild symptoms, 2 = moderate symptoms and 3 = severe symptoms
Change in patient-reported anterior rhinorrhea and posterior rhinorrhea score | From baseline to Week 24
  0-3 scale, component of patient-reported total symptom score
Change in rhinosinusitis visual analog scale (VAS). | From baseline to Week 24
  The VAS for rhinosinusitis is used to evaluate the total severity (30). Rhinosinusitis disease can be divided into Mild, Moderate and Severe based on total severity VAS score (0 to 10 cm):
  * MILD = VAS 0 to 3.
  * MODERATE = VAS >3 to 7.
  * SEVERE = VAS >7 to 10. The participant is asked to indicate along a 10 centimeter straight horizontal line (VAS) the answer to the question: "How troublesome are your symptoms of your rhinosinusitis". The VAS ranks from 0 (Not troublesome) to 10 (Worst thinkable troublesome) and is measured in centimeters.
Change in University of Pennsylvania Smell Identification Test (UPSIT) score. | From baseline to Week 24
  The UPSIT test is a rapid and easy-to-administer method to quantitatively assess human olfactory function. The test consists of four booklets, each containing 10 odorants with one odorant per page. Above each odorant strip is a multiple-choice question with four alternative words to describe the odour. Score depends on the amount of answers out of 40 possible correct answers.
Change in patient-reported loss of smell score | From baseline to Week 24
  0-3 scale, component of patient-reported total symptom score
Serum lunsekimig concentrations | From baseline to end of study (approximately 36 weeks)
Anti-drug antibodies (ADA) against lunsekimig | From baseline to end of study (approximately 36 weeks)
Incidence of participants with treatment-emergent adverse events (TEAEs) | From baseline to end of study (approximately 36 weeks)
Incidence of participants with adverse events of special interest (AESI) | From baseline to end of study (approximately 36 weeks)
Incidence of participants with serious adverse events (SAEs) | From baseline to end of study (approximately 36 weeks)
Change in asthma control questionnaire (ACQ-5) | From baseline to Week 24
  ACQ-5 is Asthma control questionnaire assessing symptoms. Lower score shows better asthma control
Change in pre-bronchodilator forced expiratory volume in the first second (pre-BD FEV1) | From baseline to Week 24
Change in pre-BD percent predicted FEV1 | From baseline to Week 24

CONTACTS AND LOCATIONS:
Locations (29):
- United States (14):
  - Allergy & Rheumatology- Site Number : 8400005, La Jolla, California
  - Sacramento Ear Nose & Throat - Roseville- Site Number : 8400003, Roseville, California
  - Senta Clinic- Site Number : 8400025, San Diego, California
  - James A Haley Veterans' Hospital- Site Number : 8400015, Tampa, Florida
  - Emory University Hospital Midtown- Site Number : 8400012, Atlanta, Georgia
  - The Allergy Group - Asthma & Allergy Boise- Site Number : 8400002, Boise, Idaho
  - Harvard Medical School - Brigham and Women's Hospital Site Number : 8400016, Boston, Massachusetts
  - Essential Medical Research- Site Number : 8400020, Tulsa, Oklahoma
  - McGovern Medical School - UT Physicians Dermatology - Bellaire Station- Site Number : 8400017, Bellaire, Texas
  - Gary Gross Pharmaceutical Research & Consulting, Inc. Site Number : 8400004, Dallas, Texas
  - Berkson Medical - McKinney- Site Number : 8400014, McKinney, Texas
  - Alamo ENT Associates Site Number : 8400001, San Antonio, Texas
  - Advanced Research Institute - Odgen- Site Number : 8400022, Ogden, Utah
  - Eastern Virginia Medical School (EVMS) Medical Group- Site Number : 8400008, Norfolk, Virginia
- Argentina (3):
  - Investigational Site Number : 0320002, Rosario, Santa Fe Province
  - Investigational Site Number : 0320001, Buenos Aires
  - Investigational Site Number : 0320003, Mendoza
- Belgium (2):
  - Investigational Site Number : 0560002, Ghent
  - Investigational Site Number : 0560001, Leuven
- Investigational Site Number : 1000001, Sofia, Bulgaria
- Poland (6):
  - Investigational Site Number : 6160002, Krakow, Lesser Poland Voivodeship
  - Investigational Site Number : 6160001, Warsaw, Masovian Voivodeship
  - Investigational Site Number : 6160005, Warsaw, Masovian Voivodeship
  - Investigational Site Number : 6160003, Katowice, Silesian Voivodeship
  - Investigational Site Number : 6160004, Poznan
  - Investigational Site Number : 6160007, Wroclaw
- United Kingdom (3):
  - Investigational Site Number : 8260004, Gloucester, Gloucestershire
  - Investigational Site Number : 8260003, Manchester
  - Investigational Site Number : 8260001, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: Chronic Rhinosinusitis with Nasal Polyps — https://www.sanofistudies.com/FGE2/
- See also: ACT18207 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=25761&tenant=MT_SNY_9011